CLINICAL TRIAL: NCT05188573
Title: EpiDetect Study: Clinical Validation of a Pancreatic Cancer Detection Test in New-Onset Diabetes Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ClearNote Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: EpiDetect
Record Dates: First submitted 2021-12-27; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; Early pancreatic cancer detection
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- EpiDetect Arm (Experimental): Each subject can undergo to up to 3 blood draws; at the time of enrollment (T0), at 6 months (T1) and 12 months (T2) from diabetes diagnosis. After 24 months from diabetes diagnosis, a review of the electronic medical records (EMR) will be performed for all subjects with a "not detected" test result.
  Interventions: Device: Early detection pancreatic cancer test
- EpiDetect "not detected" MRI Arm (Experimental): A pre-specified number of cases with test results "not detected" will be randomly selected, gender ratio and age matched to subjects with test results "detected" and will undergo MRI imaging at T0 (n=226), at T1 (n=208 ) at T2 (n=208 ) and 24 months (n=208) from diabetes diagnosis.
  Interventions: Device: Early detection pancreatic cancer test and MRI Imaging

INTERVENTIONS:
Device: Early detection pancreatic cancer test — Blood collection and pancreatic cancer early detection testing with return of results
  Arms: EpiDetect Arm
Device: Early detection pancreatic cancer test and MRI Imaging — Blood collection and pancreatic cancer early detection testing with return of results and MRI Imaging
  Arms: EpiDetect "not detected" MRI Arm

SUMMARY:
Bluestar Genomics has developed a non-invasive test that aids in the qualitative detection of occult pancreatic cancer in patients with new onset type II diabetes (NOD) who are 50 years old or older. The purpose of this study is to validate the performance of Bluestar Genomics early-detection pancreatic cancer test. The study is prospective, longitudinal and interventional; tests will be ordered and results returned to site-investigators. If the assay returns a pancreatic cancer signal "detected" result, the study participant will undergo MRI imaging to evaluate for the presence of pancreatic cancer. The study is planned to enroll 10,000 newly diagnosed type II diabetic subjects according to inclusion and exclusion criteria.

DETAILED DESCRIPTION:
This is a prospective longitudinal and interventional study of the Bluestar Genomics early detection pancreatic cancer test. The test will be ordered and results returned to site-investigators. The study is planned to enroll 10,000 male and female, ≥ 50 years of age and newly diagnosed with type II diabetes (within 90 days prior to enrollment). The study population will target 70% of subjects over 65 years old, 53% males and will target to enroll at least 50% of subjects with a BMI <32.

Each subject can undergo to up to 3 blood draws; at the time of enrollment (T0), at 6 months (T1) and 12 months (T2) from diabetes diagnosis. If test result is "detected", MRI imaging will be performed to further assess the pancreas. If the MRI imaging study results are abnormal, the subject will be referred back to their enrolling clinician for additional diagnostic work up as part of routine healthcare. After 24 months from diabetes diagnosis, a review of the electronic medical records (EMR) will be performed for all subjects with a "not detected" test result.

The study will also include an Bluestar Genomics's test "not detected" imaging arm (negative control imaging arm) for each time point. Subjects included in the negative imaging arm will be pre-specified and randomly selected among the Bluestar Genomics "not detected" cases gender ratio and age matched to Bluestar Genomics "detected" and will undergo MRI imaging.

ELIGIBILITY:
Inclusion Criteria:

* ≥50 years of age or older at the time of enrollment
* Willing to provide and sign the informed consent form
* Must have 2 occurrences from among the below parameters of diabetes mellitus (PDMs) in past 90 days measured in outpatient setting (not in urgent care, emergency room or while inpatient):
* FBG ≥126mg/dl
* HbA1c ≥ 6.5%
* RBG ≥200mg/dl
* 2-hour post-glucose ≥ 200mg/dl (OGTT)
* Must have had glycemic parameter measured in 3-18 months prior to screening without meeting DM criteria
* Must be willing to provide several tubes of blood without endangering health
* No history of pancreatic cancer
* No history of IPMNs, other neoplastic cysts and pancreatitis
* No active cancers within the past 5 years (with the exception of non-melanoma skin cancers resolved/treated > 1 year prior to enrollment and in situ carcinomas)

Exclusion Criteria:

* Prior DM diagnosis
* Met criteria for DM ≥91 days prior to enrollment (patients with prior gestational diabetes that has resolved are NOT acceptable to enroll)
* Carried a DM diagnosis or used anti-DM medications at a time greater than or equal to 91 days prior to enrollment
* Any known pancreatic lesions
* Received cancer treatment within the past 5 years (with the exception of treatment of non- melanoma skin cancer), carrying a current cancer diagnosis, and/or being investigated for suspicion of past cancer recurrence.
* Current chronic or acute oral steroid use
* History of intra-articular steroid injections (<1 week) of the qualifying DM blood test (allowed exception: nasal, topical, oral budesonide)
* Any surgery requiring general anesthesia within 2 months of collection
* Local anesthetic (including dental novocaine) within 1 week of collection
* History or presence of HIV/AIDs, Hepatitis A or E within the past five years, TB, any kind of prion disorder (e.g., CJD)
* Blood transfusion within 1 month
* Organ transplant recipient
* Currently pregnant, or pregnancy within last 12 months
* Receipt of systemic immunomodulation therapy within past 12 months
* Significant medical condition that in the site investigator's opinion would compromise the subject's ability to tolerate study interventions

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Clinical performance of test: pancreatic cancer sensitivity | 24 months or until diagnostic resolution
  Test sensitivity (Sn) for histopathology confirmed pancreatic cancer (ground truth)
Clinical performance of test: IPMNs sensitivity | 24 months or until diagnostic resolution
  Test sensitivity (Sn) for intraductal papillary mucinous neoplasms (IPMNs)
Clinical performance of test: Specificity | 24 months or until diagnostic resolution
  Test specificity (Sp) for pancreatic neoplasia.

SECONDARY OUTCOMES:
Positive Predictive Value | 24 months or until diagnostic resolution
  PPV for pancreatic neoplasia
Negative Predictive Value | 24 months or until diagnostic resolution
  NPV
Stage Shift | 24 months or until diagnostic resolution
  Evaluation of stage at diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Bethel, MD, Principal Investigator — Bluestar Genomics
Locations (1):
- Bluestar Genomics, Inc., San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No